CLINICAL TRIAL: NCT04369456
Title: Blood Innate Biomarkers as Predictors of COVID-19 Disease Progression in Recently Infected Kidney Transplant Patients
Brief Title: Blood Biomarkers as Predictors of COVID-19 Disease Progression in Recently Infected Kidney Transplant Patients
Acronym: PredictCovidT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-PP-09
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplant; Complications; Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 kidney transplant patients with moderate symptoms (Other)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — a blood sample is taken on Covid-19 kidney transplant patients with moderate symptoms

SUMMARY:
SARS-CoV-2 induces over-production of inflammatory cytokines, and especially interleukin-6 (IL-6). The apparently strong association between blood levels of inflammaory cytokines and SARS-CoV-2 disease severity has led clinicians to evaluate the administration of steroids or anti-IL-6 antagonists in severely ill patients. As of this day, biomarkers capable of predicting clinical disease progression in Covid-19 patients with mild-to-moderate symptoms have not yet been formally identified. Identifying such markers and evaluating their predictive value may be exploited to guide patient care management, and as such forms the core objective of this proposal.

Because of strong inter-individual variations in the ability of innate immune cells to produce cytokines, the hypothesis formulate and intend to test is that innate IL-6 responsiveness varies between recently infected Covid-19 patients and could predict disease outcome.

To test this hypothesis, the investigator propose to follow recently infected kidney transplant patients with moderate Covid-19 symptoms. These patients stand a higher risk to progress to severe disease. The staff plan to collect a blood sample in these patients using a system whereby ex vivo cytokine production is initiated in the very same blood collection tube without prior separation and centrifugation, thus reducing labour and operator bias. After incubation with or without known innate immune stimuli, the cell-free phase from each collection-culture tube will be assayed for IL-6 content. Associations between IL-6 content and disease outcome (encephalopathy, transfer to acute care or death) will be determined in 115 Covid-19 kidney transplant patients with moderate symptoms followed in 9 centers.

ELIGIBILITY:
Inclusion Criteria:

* Kidney or kidney-pancreas or kidney-heart transplant patients;
* SARS-CoV-2 positive (RT-PCR);
* COVID-19 symptoms at least once over a 8-day period preceding inclusion;
* Hospitalized or outpatients in one of the study centers: CHU de Nice, CHU de Strasbourg, Hôpital Necker (APHP), Hôpital Kremlin Bicêtre (APHP), Hôpital Pitié-Salpétriêre (APHP), Hospices Civils de Lyon, CHU de Saint-Etienne, CHU de Montpellier, Hôpital La Conception (APHM);
* Age > 18 years;
* Free and informed consent.

Exclusion Criteria:

* Age > 85 years ;
* Kidney-liver transplant patients;
* Onset of symptoms (fever and/or cough) for more than 8 days;
* Acute respiraytory distress despite oxygen therapy, 02 ≥ 4L/min, arterial pressure < 85/55 mmHg or hemodynamic instability at time of inclusion, encephalopathy with Glasgow coma scale < 14;
* Treatment with non-steroids anti-inflammatory agents within the last 14 days preceding onset of symptoms;
* Active bacterial or fungal infection documented at inclusion;
* Pregnancy;
* Under guardianship or curatorship;
* Non-affiliated person with Social Security

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Predictive value of IL-6 contents of whole blood samples after ex vivo stimulation | 10 months
  quantity of IL-6 in of whole blood samples after ex vivo co-stimulation with LPS and ATP in Covid-19 kidney transplant patients.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Lyon Univerity Hospital, Lyon
  - APHM, Marseille
  - Montpellier University Hospital, Montpellier
  - University Nice Hospital, Nice
  - APHP, Paris
  - Saint Etienne University Hospital, Saint-Etienne
  - Strasbourg Univeristy Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No